CLINICAL TRIAL: NCT07212036
Title: The Utilization of Ultrasound to Diagnose Pediatric Elbow Fractures: Evaluation of Cost Savings, Radiation Exposure, and Patient Satisfaction
Brief Title: The Utilization of Ultrasound to Diagnose Pediatric Elbow Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Jason Malone, Pediatric Orthopedic Surgeon, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2051060
Record Dates: First submitted 2025-09-08; First posted 2025-10-21 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Elbow Pain; Supracondylar Humerus Fracture; Radial Head Fractures; Radial Head or Neck Fractures; Elbow Dislocation; Humerus Fractures; Jakob II Classification
Keywords: elbow pain; elbow fracture; supracondylar humerus fracture; pediatric; lateral humeral condyle fracture; radial head fracture; radial neck fracture; monteggia fracture; elbow dislocation; radial head dislocation; emergency department; ultrasound
MeSH Terms: conditions — Radial Head and Neck Fractures; Humeral Fractures; Elbow Fractures; Monteggia's Fracture; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Patients elbow pain diagnosed with ultrasound (Experimental): Patients with elbow pain will receive an ultrasound of the elbow to evaluate for the present of an elbow fractures, hemarthrosis and/or lipohemarthrosis
  Interventions: Diagnostic Test: Ultrasound of the elbow
- Patient elbow pain diagnosed with x-ray (Active Comparator): Patients with elbow pain will review a standard two view elbow x-ray (anterior- posterior and lateral) to evaluate for a fracture around the elbow and/or hemarthrosis.
  Interventions: Diagnostic Test: X-ray of elbow

INTERVENTIONS:
Diagnostic Test: Ultrasound of the elbow — An ultrasound of the elbow obtained of pediatric patients with elbow pain
  Arms: Patients elbow pain diagnosed with ultrasound
Diagnostic Test: X-ray of elbow — An x-ray of the elbow obtained of pediatric patients with elbow pain
  Arms: Patient elbow pain diagnosed with x-ray

SUMMARY:
The goal of this intervention trial is to learn if a ultrasound diagnosis of elbow fractures can improve care in pediatric patients seen in the emergency room. The main questions it aims to answer are:

The primary outcomes measured are cost of the emergency visit, radiation exposure, time spent in the emergency department and patient satisfaction.

Patients who are evaluated with ultrasounds of the elbow will be compared to patients who have x-rays of the elbow.

Participants will be assigned either to the ultrasound group or x-rays group when they present with elbow pain.

DETAILED DESCRIPTION:
The goal of this study is to evaluate whether the use of point-of-care ultrasonography (PoCUS) for elbow trauma evaluation results in less radiation exposure, less cost of treatment and shorter length of stay in Emergency Room (ER) than use of radiography. The study team will use PoCUS to screen for isolated elbow fractures presented to the ER. The researchers will compare cost of treatment both for patients and health care system and length of stay in both the groups. This study will also evaluate whether the use of PoCUS alleviates discomfort to pediatric patients and increases satisfaction of the families as compared to the use of radiography. Family satisfaction surveys and patient pain surveys will act as direct measures of family satisfaction. The study team will use length of stay and cost of treatment as indirect measures of satisfaction. The researchers will compare amount of comfort and satisfaction with and without the use of PoCUS to evaluate the overall patient comfortability and patient satisfaction. The researchers hypothesize that the use of PoCUS will reduce time of emergency department length of stay, radiation exposure, pain or discomfort and cost, and will increase patient's and family satisfaction.

ELIGIBILITY:
Inclusion Criteria:

• Pediatric patient with elbow pain

Exclusion Criteria:

* Polytrauma (more than one injury)
* Deformity of the arm including the elbow
* Pain in any other location than the elbow
* Pain in other parts of the same limb including the, wrist, forearm, shoulder, hand
* Pain in other limbs,
* Puckering of the skin (skin indentation)
* Obvious fracture
* Open wound at or around the elbow
* Pain and swelling without trauma
* Concerns for tumor or infection
* Suspected nursemaid's elbow

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 225 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-02 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | Day 1
  The patient satisfaction scores will be collected by the research assistant using the Emergency Department Consumer Assessment of Healthcare Providers and Systems Survey (ED CAHPS Survey) Version 1.0. The survey will be scored based on the recommended guidelines from CAHPS. Please see the attached scoring guidelines for further information.
cost of treatment | Day 1
  Cost of treatment: will be based from hospital charges in United States Dollars (USD). The cost will be based off the cash charge for the 3-4 view x-rays of the elbow. This information is readily available online and is currently $652.00
  . It would be impossible to base from reimbursement as each insurance provider reimburses at a different rate. No cost will be assigned for the ultrasound as it is a point of care (POC) device that has no charge.

SECONDARY OUTCOMES:
Length of Stay | Day1
  calculated and recorded in EPIC. The time in minutes will be calculated from from the start when the patient is registered in the ED. All patients are registered and triaged when they enter the ED lobby. The time in ED in Epic is then stopped when the patient is discharged by the nurse.
Pain During Imaging Procedure | Day 1
  Patient pain scores who are younger than 3 years will be collected by using The FLACC score (for face, legs, activity, cry, concealability) The pain scores will be collected using the Wong-Baker FACES Pain Rating Scale for patients ages equal to and greater than 3 years old.

CONTACTS AND LOCATIONS:
Overall Officials: Jason B Malone, DO, Principal Investigator — Nemours Children's Health
Locations (1):
- Nemours Children's Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beaumont WH. Additives in feed and the E.E.C. Vet Rec. 1973 Jan 27;92(4):103. doi: 10.1136/vr.92.4.103-a. No abstract available. PMID 4693383
- [Background] Brogan M, Chakeres DW. Computed tomography and magnetic resonance imaging of the normal anatomy of the temporal bone. Semin Ultrasound CT MR. 1989 Jun;10(3):178-94. PMID 2697336
- [Background] Hall EJ. Lessons we have learned from our children: cancer risks from diagnostic radiology. Pediatr Radiol. 2002 Oct;32(10):700-6. doi: 10.1007/s00247-002-0774-8. Epub 2002 Jul 19. PMID 12244457
- [Background] Avci M, Kozaci N, Beydilli I, Yilmaz F, Eden AO, Turhan S. The comparison of bedside point-of-care ultrasound and computed tomography in elbow injuries. Am J Emerg Med. 2016 Nov;34(11):2186-2190. doi: 10.1016/j.ajem.2016.08.054. Epub 2016 Aug 27. PMID 27645809
- [Background] Lee SH, Yun SJ. Diagnostic Performance of Ultrasonography for Detection of Pediatric Elbow Fracture: A Meta-analysis. Ann Emerg Med. 2019 Oct;74(4):493-502. doi: 10.1016/j.annemergmed.2019.03.009. Epub 2019 May 9. PMID 31080032
- [Background] Mettler FA Jr, Huda W, Yoshizumi TT, Mahesh M. Effective doses in radiology and diagnostic nuclear medicine: a catalog. Radiology. 2008 Jul;248(1):254-63. doi: 10.1148/radiol.2481071451. PMID 18566177
- [Background] Burnier M, Buisson G, Ricard A, Cunin V, Pracros JP, Chotel F. Diagnostic value of ultrasonography in elbow trauma in children: Prospective study of 34 cases. Orthop Traumatol Surg Res. 2016 Nov;102(7):839-843. doi: 10.1016/j.otsr.2016.07.009. Epub 2016 Sep 30. PMID 27697406
- [Background] Eckert K, Ackermann O, Janssen N, Schweiger B, Radeloff E, Liedgens P. Accuracy of the sonographic fat pad sign for primary screening of pediatric elbow fractures: a preliminary study. J Med Ultrason (2001). 2014 Oct;41(4):473-80. doi: 10.1007/s10396-014-0525-0. Epub 2014 Mar 6. PMID 27278028
- [Background] Rabiner JE, Khine H, Avner JR, Friedman LM, Tsung JW. Accuracy of point-of-care ultrasonography for diagnosis of elbow fractures in children. Ann Emerg Med. 2013 Jan;61(1):9-17. doi: 10.1016/j.annemergmed.2012.07.112. Epub 2012 Nov 9. PMID 23142008
- [Background] Kraus R, Berthold LD, von Laer L. [Efficient imaging of elbow injuries in children and adolescents]. Klin Padiatr. 2007 Sep-Oct;219(5):282-7. doi: 10.1055/s-2007-970588. German. PMID 17763294
- [Background] Crowther M. Elbow pain in pediatrics. Curr Rev Musculoskelet Med. 2009 Jun;2(2):83-7. doi: 10.1007/s12178-009-9049-4. Epub 2009 Mar 14. PMID 19468873

DOCUMENTS (5):
  • Study Protocol and Statistical Analysis Plan (2025-03-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT07212036/Prot_SAP_005.pdf
  • Informed Consent Form: Seven to Eleven Year old Assent (2025-05-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT07212036/ICF_001.pdf
  • Informed Consent Form: Parental Permission (2025-05-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT07212036/ICF_002.pdf
  • Informed Consent Form: Informed Consent (2025-05-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT07212036/ICF_003.pdf
  • Informed Consent Form: Children's Assent 12-17 years old (2025-05-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT07212036/ICF_004.pdf